CLINICAL TRIAL: NCT05337644
Title: Leak After Sleeve Gastrectomy With Positive Intraoperative Indocyanine Green Test: Avoidable Scenario?
Brief Title: Indocyanine Green Test for Evaluation of Perfusion of Staple Line of the Stomach During Laparoscopic Sleeve Gastrectomy
Status: Completed | Type: Observational
Sponsor: University of Foggia (Other)
Responsible Party: Principal Investigator, Giovanna Pavone, Medical doctor, University of Foggia
Other Study IDs: 4
Record Dates: First submitted 2022-03-30; First posted 2022-04-20 (Actual); Last update posted 2022-04-20 (Actual); Status verified 2022-04

CONDITIONS: Obesity, Morbid; Diabete Type 2; Cardiac Disease; Vascular Diseases
Keywords: laparoscopic Sleeve gastrectomy; Bariatric Surgery; Indocyanine greene test; gastric fistula
MeSH Terms: conditions — Obesity, Morbid; Diabetes Mellitus, Type 2; Heart Diseases; Vascular Diseases; Gastric Fistula

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

INTERVENTIONS:
Drug: Indocyanine green solution — 5 ml of ICG were then injected intravenously to identify the stomach, carefully assessing the angle of His (preoperative written informed consent was obtained from the patient).
  Adequate perfusion was defined as "the direct and clear visualization of the fluorescence around the gastric tube, after an estimated time of 150-180 s followingi.v. administration".

SUMMARY:
The investigators present the case of a 40-year-old female underwent laparoscopic sleeve gastrectomy. Intraoperative indocyanine green test was performed

ELIGIBILITY:
Inclusion Criteria:

* BMI >40 kg/m2

Exclusion Criteria:

* Non-obese patients

Ages: 18 Years to 65 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Obese patients with BMI >40 kg/m2 underwent laparoscopic Sleeve gastrectomy
Sampling Method: Probability Sample
Enrollment: 1 (Actual)
Dates: Start 2022-01-21 (Actual); Primary Completion 2022-02-06 (Actual); Study Completion 2022-03-25 (Actual)

PRIMARY OUTCOMES:
Positive Intraoperative Indocyanine green test | from 20 January 2022 to 20 January 2022
  Intraoperative indocyanine green test was performed

CONTACTS AND LOCATIONS:
Overall Officials: Antonio Ambrosi, Study Chair — University of Foggia
Locations (1):
- University of Foggia, Foggia, Italy

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Pavone G, Tartaglia N, Pacilli M, Maddalena F, Petruzzelli F, Ambrosi A. Leak after sleeve gastrectomy with positive intraoperative indocyanine green test: Avoidable scenario? Int J Surg Case Rep. 2022 Jun;95:107168. doi: 10.1016/j.ijscr.2022.107168. Epub 2022 May 6. PMID 35567877

DOCUMENTS (1):
  • Study Protocol (2022-03-30): https://cdn.clinicaltrials.gov/large-docs/44/NCT05337644/Prot_000.pdf